CLINICAL TRIAL: NCT04571138
Title: Pediatric and Young Adult Leukemia Adoptive Therapy (PLAT)-07: A Phase 1/2 Study of CD22-Specific CAR T Cells for CD22+ Leukemia or Lymphoma
Brief Title: A Pediatric and Young Adult Trial of Genetically Modified T Cells Directed Against CD22 for Relapsed/Refractory Leukemia or Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Colleen Annesley, Medical Director, Seattle Children's Therapeutics, Seattle Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLAT-07
Record Dates: First submitted 2020-09-02; First posted 2020-09-30 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-04

CONDITIONS: Leukemia; Lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- SCRI-CAR22v2 (Experimental): Patients will receive SCRI-CAR22v2 in either Phase I or Phase II
  Interventions: Biological: SCRI-CAR22v2

INTERVENTIONS:
Biological: SCRI-CAR22v2 — Single infusion of SCRI-CAR22v2

SUMMARY:
Patients with relapsed or refractory leukemia or lymphoma are often refractory to further chemotherapy. In this study, the investigators will attempt to use T cells obtained directly from the patient, which can be genetically engineered to express a chimeric antigen receptor (CAR). The CAR used in this study can recognize CD22, a protein expressed on the surface of leukemia and lymphoma cells. The phase 1 part of this study will determine the safety and appropriate dose level of these CAR T cells, and the phase 2 part of the study will determine how effective this CAR T cell therapy is. Both patients who have never had prior CAR T cell therapy and those who have had prior CAR T cell therapy may be eligible to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged ≤ 30 years. First 2 enrolled subjects: age ≥ 18 and ≤ 30 years
* Evidence of refractory or recurrent CD22+ leukemia or lymphoma
* Able to tolerate apheresis, or subject with sufficient existing apheresis product or T cells for manufacturing investigational product.
* Life expectancy ≥ 8 weeks
* Lansky or Karnofsky, as applicable, score ≥ 50
* Recovered from acute toxic effects of all prior chemotherapy, immunotherapy, and radiotherapy, if the subject does not have a previously obtained apheresis product that is acceptable and available for manufacturing of CAR T cells
* ≥ 7 days post last chemotherapy and biologic therapy, with the exception of intrathecal chemotherapy and maintenance chemotherapy
* ≥ 7 days post last corticosteroid therapy
* ≥ 3 days post Tyrosine Kinase Inhibitor (TKI) use
* ≥ 1 day post hydroxyurea
* 30 days post most recent CAR T cell infusion
* Adequate organ function
* Adequate laboratory values, including absolute lymphocyte count ≥ 100 cells/uL
* Subjects of childbearing or child-fathering potential must agree to use highly effective contraception from consent through 12 months following infusion of investigational product on trial
* Subject and/or legally authorized representative has signed the informed consent form for this study

Exclusion Criteria:

* Presence of active malignancy other than disease under study
* History of symptomatic CNS pathology or ongoing symptomatic CNS pathology
* CNS involvement of leukemia or lymphoma that is symptomatic and in the opinion of the investigator, cannot be controlled during the interval between enrollment and CAR T cell infusion
* Subjects with uniform expression of CD19 on their malignant cells who are eligible but have not attempted CD19 directed CAR T cell therapy
* For subjects having had a previous stem cell transplant: presence of active GVHD, or receiving immunosuppressive therapy for treatment or prevention of GVHD within 4 weeks prior to enrollment
* Presence of active severe infection,
* Presence of primary immunodeficiency syndrome
* Subject has received prior virotherapy
* Pregnant or breastfeeding
* Subject and/or legally authorized representative unwilling to provide consent/assent for participation in the 15-year follow-up period, required if CAR T cell therapy is administered
* Presence of any condition that, in the opinion of the investigator, would prohibit the subject from undergoing treatment under this protocol

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Estimated)
Dates: Start 2020-09-25 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2040-02 (Estimated)

PRIMARY OUTCOMES:
The adverse events associated with CAR T cell product infusions will be assessed | 28 days post-infusion
  The type, frequency, severity, and duration of adverse events will be summarized
The ability to successfully manufacture SCRI-CAR22v2 | 28 days
  We will measure the number of successfully manufactured SCRI-CAR22v2 products
The leukemia response to SCRI-CAR22v2 in subjects with relapsed or refractory CD22+ leukemia will be assessed | 28 days post-infusion
  The efficacy of the T cell infusion will be estimated based on the number of participants who have an MRD negative bone marrow aspirate following the T cell infusion

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Summers, MD, Study Chair — Seattle Children's Hospital
Locations (5):
- United States (5):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's National Hospital, Washington D.C., District of Columbia
  - Riley Hospital for Children, Indianapolis, Indiana
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No